CLINICAL TRIAL: NCT00356785
Title: Body Compositional and Endocrine-Metabolic Changes by Long-Term Lifestyle Intervention With Health Education, Diet (Almased®), Physical Activity or a Combination of Diet and Physical Activity in Overweight and Obese Persons.
Brief Title: Changes in Body Composition and Metabolic Risk Parameters by Life Style Intervention.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Almased Wellness GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 230/01
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-04

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: lifestyle; diet; exercise; physical activity; obesity
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Motor Activity | interventions — Dietary Supplements

INTERVENTIONS:
Behavioral: health education
Behavioral: food supplementation
Behavioral: food supplementation combined with physical activity program

SUMMARY:
Eligible overweight and obese persons will be randomized to one of three controlled groups: 1 group of participants is treated by health education for life style intervention only. The other 2 groups will be included in a dietary program with an individually dosed food supplement (Almased®) for an initial weight reduction for a period of 6 weeks. The following 18 weeks represent the most important phase of weight loss and attitude, the participants take part in 2 different interventions according to their randomization. One group will continue the dietary program, one group will try to achieve and maintain weight reduction by continuing the initial dietary program together with an additional physical activity program. For all intervention groups the following 6 months aim at a further stabilization of weight and attitude, now without defined guidelines of intervention but with the intention to continue the so far practiced change in life style. All participants will be supplied with adequate information and material concerning the desired change in life style.

DETAILED DESCRIPTION:
Obese and adipose participants are randomized to three intervention groups. During the first six weeks of the program, the subjects assigned to the substitutional diet group (SD-G) were instructed to replace two daily meals with a commercially available soy-joghurt-honey preparation (Almased®). During the following 18 weeks, only one daily meal was replaced by the preparation. The dietary intake of fat during this second phase was not to exceed 60g per day. The first 6-week diet contained about 1000 kcal per day for women and 1200 kcal for men, and then, in the following weeks, aimed at a maximum of 1500 kcal for women and 1700 kcal for men. In addition, a second group of subjects were encouraged to additionally attend a 60-minute physical activity endurance program twice weekly. Otherwise, they were to follow the same rules as the substitutional diet group (SD/PA-G).

The lifestyle education group (LE-G) attended, after enrolment, three teaching sessions bi-monthly and had individual consultations during weeks 6, 24 and 48. All sessions were held by experts in nutritional counselling. Subjects received a diet-overview handout, in accordance with the "German Society of Nutrition" and the "German Society of Sports Medicine and Prevention". Prescribed was a moderate-fat, nutrient-balanced reduction diet consisting of 1200 to 1500 kcal per day for women and 1500 to 1800 kcal per day for men, with approximately 60 percent of the calories coming from carbohydrates, 25 percent from fat, and 15 percent from protein.

The data collected at enrolment and after 6, 24 and 48 weeks were body weight, waist and abdominal circumference, self-reported medical history, blood pressure, glucose, insulin, serum lipids and inflammatory markers (C-reactive protein, IL-6). For measurement of body composition, the technique of air displacement plethysmography was used (Bod Pod). Dietary compliance was estimated by 24-hour recalls of dietary consumption.

Endpoints: Body weight loss of 5% and 10 %; Reduction of body fat; Change of muscle mass

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must have overweight with a BMI between 27,5 and 35 kg/m²
* The participants must be able to participate in a physical activity program
* The participants must be willing to participate in the program for 1 year
* Written informed consent must be given to accept randomization to either of the intervention groups

Exclusion Criteria:

* Participants who do not meet all entry criteria
* BMI > 35,0 kg / m²
* Performance capacity < 75 w for 2 min
* Subjects younger than 35 yrs (with reference age at 1st Jan 2002: 34.5 yrs) or older than 65 yrs (with reference age at 1st 2002: 65.5 yrs)
* Absolute or relative contraindications to exercise testing of the ACSM
* Persons unable or with restrictions to participate in a regular physical activity program because of any disease (e.g. history of CHD, arrhythmia, valvular heart disease, arthritis of major joints)
* Severe hypertension systolic BP of > 200 mm Hg and or diastolic BP of > 105 mm Hg at rest
* Persons with established insulin dependent diabetes mellitus (IDDM)
* Persons with a disease of the liver or the kidneys prohibiting high protein intake
* Persons with a disease of the thyroid gland or taking thyroid hormones

Ages: 34 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2001-01; Study Completion 2001-12

PRIMARY OUTCOMES:
body weight loss of more than 5%
body weight loss of more than 10%

SECONDARY OUTCOMES:
reduction of body fat
change of muscle mass
change in blood pressure
change in lipids
change in fasting blood glucose
change in weight circumference

CONTACTS AND LOCATIONS:
Overall Officials: Aloys Berg, Prof.Dr., Study Director — University Hospital, Department for Rehabilitation, Prevention and Sports Medicine, Freiburg, Germany
Locations (1):
- University Hospital, Department for Rehabilitation, Prevention and Sports Medicine, Freiburg im Breisgau, Germany

REFERENCES:
- [Result] Deibert P, Konig D, Schmidt-Trucksaess A, Zaenker KS, Frey I, Landmann U, Berg A. Weight loss without losing muscle mass in pre-obese and obese subjects induced by a high-soy-protein diet. Int J Obes Relat Metab Disord. 2004 Oct;28(10):1349-52. doi: 10.1038/sj.ijo.0802765. PMID 15303108
- [Derived] Koohkan S, Schaffner D, Milliron BJ, Frey I, Konig D, Deibert P, Vitolins M, Berg A. The impact of a weight reduction program with and without meal-replacement on health related quality of life in middle-aged obese females. BMC Womens Health. 2014 Mar 12;14(1):45. doi: 10.1186/1472-6874-14-45. PMID 24618460